CLINICAL TRIAL: NCT03244982
Title: Comparison of Timing and Image Quality of Different Phases of Optos Fluorescein Angiography Between Two Doses of Intravenous Fluorescein: 250mg Versus 500mg
Brief Title: Fluorescein Angiography With a Full-dose Versus a Half-dose of Intravenous Fluorescein
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Additional data may be required once preliminary data is analyzed.
Sponsor: Kresge Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 23897543
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Fluorescein Angiography
Keywords: fluorescein; angiography
MeSH Terms: interventions — Fluoresceins

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to receive either a half-dose (250mg) or a full-dose (500mg) of intravenous fluorescein prior to their angiography procedure. If they return for a second fluorescein angiography study during the proceeding four months, they will receive the dose of fluorescein (250mg or 500mg) which they did not receive during their first study. Images will be evaluated subjectively by a masked panel of retinal surgeons for image quality, and image quality will be compared between images that are full dose and images that are half dose.
Who Masked: Outcomes Assessor
Masking Description: The primary outcomes assessors will be retinal surgeons and residents, masked to the dosing of fluorescein. They will assess the subjective quality of images.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Full-Dose (Active Comparator): Participants in this arm will receive Fluorescein Na 10% Inj 500mg pushed over several seconds one time, prior to their fluorescein angiogram. If they return for a second (clinically indicated) angiogram, they will receive Fluorescein Na 10% Inj 250mg pushed over several seconds one time.
  Interventions: Drug: Fluorescein Na 10% Inj 500mg; Drug: Fluorescein Na 10% Inj 250mg
- Half-Dose (Experimental): Participants in this arm will receive Fluorescein Na 10% Inj 250mg pushed over several seconds one time, prior to their fluorescein angiogram. If they return for a second (clinically indicated) angiogram, they will receive Fluorescein Na 10% Inj 500mg pushed over several seconds one time.
  Interventions: Drug: Fluorescein Na 10% Inj 500mg; Drug: Fluorescein Na 10% Inj 250mg

INTERVENTIONS:
Drug: Fluorescein Na 10% Inj 500mg — Full-dose intravenous Fluorescein Na prior to fluorescein angiography.
  Other Names: AK-Fluor
Drug: Fluorescein Na 10% Inj 250mg — Half-dose intravenous Fluorescein Na prior to fluorescein angiography.
  Other Names: AK-Fluor

SUMMARY:
Fluorescein angiography is a common procedure used in ophthalmology to diagnose and monitor diseases of the eye. The standard dose of fluorescein dye used in fluorescein angiography is 500mg. It is common practice to give patients who have previously had an adverse reaction to fluorescein dye a half-dose, or 250mg, of fluorescein. It has been determined by our institution that anecdotally, there is no difference in image quality between the images created by a half-dose of fluorescein versus a full dose of fluorescein. Therefore, this study seeks to determine whether these doses are actually equivalent in terms of image quality. Patients who consent to participate in the study will be randomized to receive either a half or a full dose of intravenous fluorescein, and their images will be compared subjectively using a masked team of retinal surgeons and residents. We hypothesize that there will be no significant difference between the images obtained using a half-dose versus a full dose of intravenous fluorescein.

DETAILED DESCRIPTION:
Fluorescein angiography is a common procedure used in ophthalmology to diagnose and monitor diseases of the retinal and choroidal blood vessels. The most commonly seen adverse reactions to fluorescein angiography include nausea, vomiting, and urticaria. More severe reactions such as anaphylaxis are rare, occurring in only 1 of 2247 patients (0.4%) in a recent retrospective study. The standard dose of intravenous fluorescein used for fluorescein angiography is 500mg given intravenously in a 10% or 25% solution. One study from 2008 attempted to compare a 200mg dose versus a 500mg dose of intravenous fluorescein, and found that 200mg produced inferior image quality. However, the quality of the cameras used for fluorescein angiography has improved significantly in the last 10 years, and the scanning laser ophthalmoscope currently used for fluorescein angiography in our clinic (Optos) is significantly more effective than the fundus camera used in the 2008 study (Topcon). The scanning laser ophthalmoscope uses a fundamentally different imaging technique than the traditional fundus camera, with a much narrower illumination source, and has been shown to be significantly more sensitive in the detection of retinal vascular leakage.

A commonly used method for preventing adverse reactions in patients who have previously had an adverse reaction to intravenous fluorescein is to use a 250mg dose instead of the standard 500mg dose, despite the lack of evidence to this effect. In our anecdotal experience, a 250mg dose of intravenous fluorescein, used in patients whom have previously experienced an adverse reaction, has produced images of equivalent quality to the images produced using a full 500mg dose. To our knowledge, no study has compared a 500mg dose of intravenous fluorescein with a lower dose since the 2008 study previously mentioned, despite the advances in camera quality.

The study will aim to recruit a sample size of approximately 100 patients. Adult patients scheduled for fluorescein angiography at the Kresge Eye Institute will be recruited into the study by one of the study members if they meet inclusion and exclusion criteria. Once a patient has consented to participate in the study, they will be randomized to receive either a 250mg or 500mg dose of intravenous fluorescein with their fluorescein angiography procedure. All fluorescein angiograms will be done only if clinically indicated, and therefore the patient will not be placed at any increased risk by participating in this study. If a participant returns for a repeat fluorescein angiogram within the next four months, they will receive the dose (250mg or 500mg) which they did not receive with their previous angiogram. Patients who experience an adverse reaction during their first angiogram will be removed from the study in order to prevent a patient who had an adverse reaction with a half-dose from receiving a full-dose with a subsequent procedure. The photographer will adjust the image brightness settings in order to create the "best possible" image for each patient, and there will be no change between procedures with the 250mg and 500mg doses. A single camera (Optos) will be used for each patient in the study.

Data collection will be obtained from the patient, the imaging procedure, and the patient's electronic medical records at the Kresge Eye Institute. Information to be collected includes age, gender, race, visual acuity, and ophthalmologic medical history. The timing and quality of images at different phases of fluorescein angiography will be compared between 500mg and 250mg doses in each eye using objective and subjective measures. Subjective criteria will include grading of the images by a panel of masked retinal surgeons and residents. Grading will look at specific factors of a fluorescein angiography such as macula detail, macrovasculature, and microvasculature. These subjective criteria will then be used to determine whether any appreciable difference exists in the image quality between 250mg and 500mg doses of intravenous fluorescein given prior to Optos fluorescein angiography.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for fluorescein angiography at Kresge Eye Institute.

Exclusion Criteria:

* Patients with known major profusion defects on fluorescein angiography.
* Patients with prior adverse reactions to fluorescein angiography.
* Patients with significant photophobia as judged by the photographer.
* Patients with visually significant cataracts.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Subjective comparison of image quality between full-dose and half-dose fluorescein angiography performed on the same patient. | Six months.
  Participants who receive two clinically-indicated fluorescein angiography procedures within the time frame of the study will receive both doses of Fluorescein Na (250mg and 500mg). These two images will then be compared to each other in terms of image quality by a team of masked retinal surgeons.

SECONDARY OUTCOMES:
Subjective comparison of image quality between full-dose and half-dose fluorescein angiography among all patients enrolled in the study. | One month.
  All of the images obtained during the patient recruitment phase of the study will be evaluated subjectively in terms of image quality by a panel of masked retinal surgeons. The images will then be compared between patients to determine if there is a subjective difference in image quality between a 250mg and 500mg dose.

CONTACTS AND LOCATIONS:
Overall Officials: Gary W Abrams, MD, Principal Investigator — Kresge Eye Institute
Locations (1):
- Kresge Eye Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu K, Tzankova V, Li C, Sharma S. Intravenous fluorescein angiography-associated adverse reactions. Can J Ophthalmol. 2016 Oct;51(5):321-325. doi: 10.1016/j.jcjo.2016.03.015. Epub 2016 Sep 3. PMID 27769320
- [Background] Moosbrugger KA, Sheidow TG. Evaluation of the side effects and image quality during fluorescein angiography comparing 2 mL and 5 mL sodium fluorescein. Can J Ophthalmol. 2008 Oct;43(5):571-5. doi: 10.3129/i08-122. PMID 18982034
- [Background] Nicholson BP, Nigam D, Miller D, Agron E, Dalal M, Jacobs-El N, da Rocha Lima B, Cunningham D, Nussenblatt R, Sen HN. Comparison of wide-field fluorescein angiography and 9-field montage angiography in uveitis. Am J Ophthalmol. 2014 Mar;157(3):673-7. doi: 10.1016/j.ajo.2013.12.005. Epub 2013 Dec 7. PMID 24321475